CLINICAL TRIAL: NCT04165317
Title: A Phase 3, Multinational, Randomized, Open-Label, Three Parallel-Arm Study of PF-06801591, an Anti-PD-1 Antibody, in Combination With Bacillus Calmette-Guerin (BCG Induction With or Without BCG Maintenance) Versus BCG (Induction and Maintenance) in Participants With High-Risk, BCG-Naïve Non-Muscle Invasive Bladder Cancer or PF-06801591 as a Single Agent in Participants With BCG-Unresponsive NMIBC
Brief Title: A Study of Sasanlimab in People With Non-muscle Invasive Bladder Cancer
Acronym: CREST
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B8011006; CREST (Other: Alias Study Number); 2023-509089-39-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Non-muscle Invasive Bladder Cancer
Keywords: CREST; Sasanlimab; PF-06801591; Bacillus Calmette Guerin; BCG; Bladder cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms | interventions — BCG Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- PF-06801591 + BCG induction and maintenance (Experimental): PF-06801591 in combination with Bacillus Calmette Guerin(induction+maintenance).
  Interventions: Drug: PF-06801591; Drug: Bacillus Calmette-Guerin
- PF-06801591 + BCG induction only (Experimental): PF-06801591 in combination with Bacillus Calmette Guerin (induction only).
  Interventions: Drug: PF-06801591; Drug: Bacillus Calmette-Guerin
- BCG induction and maintenance (Active Comparator): Bacillus Calmette Guerin (induction and maintenance).
  Interventions: Drug: Bacillus Calmette-Guerin
- BCG Unresponsive CIS (Experimental): PF-06801591
  Interventions: Drug: PF-06801591
- BCG Unresponsive NMIBC (Experimental): PF-06801591
  Interventions: Drug: PF-06801591

INTERVENTIONS:
Drug: PF-06801591 — A monoclonal antibody (mAb) that blocks the interaction between PD-1 and PD-L1/PD-L2.
  Other Names: Sasanlimab
  Arms: BCG Unresponsive CIS; BCG Unresponsive NMIBC; PF-06801591 + BCG induction and maintenance; PF-06801591 + BCG induction only
Drug: Bacillus Calmette-Guerin — Immunotherapy treatment approved by FDA for patients with high-risk non-muscle invasive bladder cancer
  Other Names: BCG
  Arms: BCG induction and maintenance; PF-06801591 + BCG induction and maintenance; PF-06801591 + BCG induction only

SUMMARY:
The purpose of this study is to learn about the safety and effects of the study medicine (sasanlimab) in people with non-muscle invasive bladder cancer. This study is seeking participants whose bladder cancer is still in early stages, has not spread outside of the bladder, has been removed with surgery, and is high risk (Part A) or was previously treated with BCG (Bacillus Calmette Guerin), a standard treatment for bladder cancer (Part B).

In Part A (enrollment closed), each participant was assigned to one of three study treatment groups.

* One group is given sasanlimab and BCG at the study clinic.
* The second group is given sasanlimab and BCG at the study clinic. This group will receive BCG for the first six weeks only.
* The third group is given BCG only and will not receive sasanlimab.

In Part B of the study, each new participant will be assigned to a study treatment group based on the type of their bladder tumor.

- Both groups will be given sasanlimab at the study clinic.

On August 31, 2022, the Sponsor announced the discontinuation of enrollment to Part B. The decision to discontinue enrollment to Part B was not made for safety reasons.

DETAILED DESCRIPTION:
CREST: Combination of sasanlimab and alternative BCG Regimens to Evaluate outcomes with Subcutaneous anti-PD-1 Treatment

Phase 3 Design with two Cohorts. Cohort A consists of 3 study Arms (A, B and C) of BCG naive participants. Arms A and B consist of two study drugs, PF-06801591 plus BCG. Arm C consists of one study drug, BCG. Cohort B consists of B1 and B2, which test PF-06801591 and include participants who have BCG unresponsive CIS (B1) or BCG unresponsive papillary only disease (B2).

The study is designed to demonstrate that PF-06801591 plus Bacillus Calmette Guerin (BCG) (induction and maintenance periods) is superior to BCG alone (induction and maintenance periods) in prolonging event free survival (EFS) in participants with high-risk naïve non-muscle invasive bladder cancer (NMIBC) and to demonstrate that PF-06801591 plus BCG (induction period only) is superior to BCG alone (induction and maintenance periods) in prolonging EFS in participants with high-risk NMIBC. The study is also designed to estimate the CR rate of PF-06801591 alone in participants with BCG unresponsive CIS and to evaluate the EFS of PF-06801591 alone in participants with BCG unresponsive NMIBC.

On August 31, 2022, the Sponsor announced the discontinuation of enrollment to Part B, which enrolled participants with BCG unresponsive NMIBC. The decision to discontinue enrollment to Part B was not made for safety reasons.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed diagnosis of high risk non-muscle invasive transitional cell carcinoma (TCC) of the urothelium of the urinary bladder (tumors of mixed transitional/non-transitional cell histology are allowed, but TCC must be the predominant histology)
* Complete resection of all Ta/T1 papillary disease (including participants with concurrent CIS), with most recent positive TURBT occurring within 12 weeks prior to randomization or study intervention. A second TURBT must have been performed if indicated according to the current locally applicable guidelines, ie, American Urological Association, European Association of Urology
* (Cohorts B1 and B2 only): Histological confirmed diagnosis of BCG-unresponsive high-risk, non-muscle invasive TCC of the urothelium within 12 months (CIS only) or 6 months (recurrent Ta/T1 disease) of completion of adequate BCG therapy.
* Have refused or are ineligible for radical cystectomy

Exclusion Criteria:

* Evidence of muscle-invasive, locally advanced or metastatic urothelial cancer or concurrent extravesical, non-muscle invasive TCC of the urothelium
* (Cohort A only): Intravesical BCG therapy within 2 years prior to randomization. Prior intravesical chemotherapy for NMIBC is allowed.

(Cohorts B1 and B2 only): Any systemic or intravesical chemotherapy or immunotherapy from the time of most recent positive TURBT to initiation of study intervention.

* Prior immunotherapy with anti PD-1, anti PD-L1, anti PD-L2, or anti cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody
* Prior treatment with immunostimulatory agents including interleukin (IL)-2, IL-15, interferon (INF)
* Prior radiation therapy to the bladder
* (Cohorts B1 and B2 only): Prior participation in Cohort A of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1068 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2026-12-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (191):
- United States (43):
  - Arizona Urology Specialists, Tucson, Arizona
  - Arkansas Urology, Little Rock, Arkansas
  - Koman Family Outpatient Pavilion, La Jolla, California
  - Sulpizio Cardiovascular Center at UC San Diego Health, La Jolla, California
  - UC San Diego Medical Center - La Jolla (Jacobs Medical Center / Thornton Pavilion), La Jolla, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of California Irvine Medical Center, Orange, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - The Urology Center of Colorado, Denver, Colorado
  - Urological Research Network Corp, Hialeah, Florida
  - UF Health Jacksonville, Jacksonville, Florida
  - UF Health North, Jacksonville, Florida
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - DuPage Medical Group, Lisle, Illinois
  - DuPage Medical Group Ambulatory Surgery Center, Lombard, Illinois
  - DuPage Medical Group, Lombard, Illinois
  - Edward Hospital, Naperville, Illinois
  - Ochsner LSU Health Shreveport - Regional Urology, Shreveport, Louisiana
  - Chesapeake Urology Research Associates, Hanover, Maryland
  - Michigan Institute of Urology, PC, Troy, Michigan
  - Bellevue Hospital, New York, New York
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - NYU Langone Medical Center (Tisch Hospital), New York, New York
  - NYU Langone Health Urology Associates, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Premier Medical Group of the Hudson Valley PC, Poughkeepsie, New York
  - Associated Medical Professionals of New York, PLLC, Syracuse, New York
  - Montefiore Medical Center - Montefiore Medical Park, The Bronx, New York
  - Montefiore Medical Center - Oncology Investigational Services, The Bronx, New York
  - VA Portland Healthcare System, Portland, Oregon
  - AUC Urologists LLC, Murrells Inlet, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Parkway Surgery Center, Myrtle Beach, South Carolina
  - Atlantic Urology Clinics South Strand Office, Myrtle Beach, South Carolina
  - Urology Clinics of North Texas, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Houston Metro Urology, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Urology San Antonio PA, San Antonio, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Chesapeake Regional Surgery Center - Virginia Beach, Virginia Beach, Virginia
  - Urology of Virginia, PLLC, Virginia Beach, Virginia
- Australia (5):
  - Southern Highlands Cancer Centre, Bowral, New South Wales
  - Chris O'Brien Lifehouse Hospital, Camperdown, New South Wales
  - Box Hill Hospital, Box Hill, Victoria
  - Eastern Clinical Research Unit, Box Hill, Victoria
  - Yarra Ranges Health, Lilydale, Victoria
- UZ Gent, Ghent, Belgium
- Canada (13):
  - Vancouver Prostate Centre at the Vancouver General Hospital, Vancouver, British Columbia
  - Hamilton Regional Laboratory Medicine Program, Hamilton, Ontario
  - Kingston Health Sciences Center - Queen's University, Kingston, Ontario
  - Centre for Applied Urological Research, Kingston, Ontario
  - Kingston Health Sciences Centre -- Hotel Dieu Hospital, Kingston, Ontario
  - University Health Network , Toronto General Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - University Health Network - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre integre universitaire de sante et de services sociaux (CIUSSS) du Saguenay-Lac-Saint-Jean, Chicoutimi, Quebec
  - Centre intégré universitaire de santé et de services sociaux (CIUSSS) du Saguenay-Lac-Saint-Jean, Chicoutimi, Quebec
  - The Research Institute of the McGill University Health Centre, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Hotel-Dieu de Quebec - CHU de Quebec - Universite Laval, Québec, Quebec
- China (21):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Chao-yang Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Affiliated First Hospital, Fuzhou, Fujian
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - Second Affiliated Hospital of Suzhou University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Chongqing University Cancer Hospital, Chongqing
  - Fudan University Cancer Hospital, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - The Second Hospital of Tianjin Medical University, Tianjin
- France (12):
  - Hôpital privé Antony (Pharmacy), Antony
  - Clinique Belharra, Bayonne
  - CHU de Bordeaux Hôpital Pellegrin, Bordeaux
  - Clinique Saint-Augustin, Bordeaux
  - Institut Bergonié, Bordeaux
  - Cabinet Privé d'urologie, Brest
  - CHPB Keraudren, Brest
  - Groupe Vivalto Sante - Clinique Pasteur-Lanroze- CFRO, Brest
  - Polyclinique de Limoges Site Chenieux, Limoges
  - Polyclinique de Gentilly, Nancy
  - Hôpital Bichat - Claude-Bernard, Paris
  - Clinique Sainte Anne, Strasbourg
- Germany (5):
  - Urologicum Duisburg, Duisburg
  - Klinikum der Goethe-Universitaet Frankfurt, Frankfurt
  - Universitaetsklinikum Muenster, Urologie, Münster
  - Studienpraxis Urologie, Nürtingen
  - Universitaetsklinikum Tuebingen, Tübingen
- Italy (16):
  - Humanitas Istituto Clinico Catanese S.p.A - U.O. Oncologia Medica, Misterobianco (CT), Catania
  - UO Oncologia, ASST di Cremona - Istituti Ospitalieri - Ospedale di Cremona, Cremona, CR
  - IRCSS Istituto Clinico Humanitas - U.O. Oncologia Medica, Rozzano, Milano
  - Ordine Mauriziano Umberto I Hospital,, Turin, Other
  - Azienda USL IRCCS di Reggio Emilia, Reggio Emilia, RE
  - Azienda Unita Sanitaria Locale Toscana Sud-Est, Arezzo
  - Ospedale Area Aretina Nord - UOC Oncologia Medica, Arezzo
  - Ospedale San Donato, Arezzo
  - UO Oncologia Medica IRCCS Istituto Tumori "Giovanni Paolo II", Bari
  - IRCCS Azienda Ospedaliera Universitaria Policlinico San Martino Urologia, Genova
  - Ospedale Generale Provinciale di Macerata - UOC Oncologia, Macerata
  - Medical Oncology Unit, AO Papardo, Messina
  - IRCCS Ospedale San Raffaele, URI (Urological Research Institute), Milan
  - AUSL/IRCCS di Reggio Emilia, Reggio Emilia
  - AO Azienda Ospedaliera Ordine Mauriziano Di Torino, Turin
  - ASST Sette Laghi Ospedale di Circolo Fondazione Macchi, Varese
- Japan (14):
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Ehime University Hospital, Tōon, Ehime
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Gunma Prefectural Cancer Center, Ōta, Gunma
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Kanagawa cancer center, Yokohama, Kanagawa
  - Osaka International Cancer Institute, Osaka, Osaka
  - Kindai University Hospital, Sayama, Osaka
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Kagoshima University Hospital, Kagoshima
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Okayama Medical Center, Okayama
  - Yamagata University Hospital, Yamagata
- Poland (10):
  - NZOZ AKMED Andrzej Kupilas, Gliwice
  - Regionalny Szpital Specjalistyczny im. Dr. Wladyslawa Bieganskiego, Grudziądz
  - Niepubliczny Zaklad Opieki Zdrowotnej Centrum Urologiczne Sp. z o.o., Mysłowice
  - Provita Profamilia, Piotrkow Trybunalski
  - Clinical Research Center Spolka z ograniczona odpowiedzialnoscia MEDIC-R Spolka Komandytowa, Poznan
  - ETG Skierniewice, Skierniewice
  - Provita 001, Warsaw
  - Medical Concierge Centrum Medyczne, Warsaw
  - Lexmedica, Wroclaw
  - Wojewódzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Łodzi, Łódż, Łódź Voivodeship
- Russia (21):
  - A.Tsyb Medical Research Radiological Center of the Ministry of Health of the Russian Federation, Obninsk, Kaluzhskaya OBL.
  - State Budgetary Institution of Healthcare of the Republic of Mordovia, Saransk, Respublika Mordoviya
  - Private Medical Institution "Euromedservice", Pushkin, Sankt-Peterburg
  - Klinika UZI 4D, LLC, Pyatigorsk, Stavropolskiy KRAI
  - Evimed Llc, Chelyabinsk
  - Regional Budgetary Healthcare Institution "Ivanovo Regional Oncology Dispensary", Ivanovo
  - Ars Medika Center, LLC, Kaliningrad
  - Kaluga Regional Clinical Oncology Center, Kaluga
  - P.A. Hertsen Moscow Oncology Research Center- branch of the National Medical Research, Moscow
  - Federal Budgetary Institution of Healthcare "Privolzhsky District Medical Center of the Federal, Nizhny Novgorod
  - National Medical Research Radiological Centre of the MoH of the Russian Federation, Obninsk
  - BHI of Omsk region "Clinical Oncological Dispensary", Omsk
  - State Budgetary Institution of Ryazan Region "Regional Clinical Oncology Center", Ryazan
  - Federal State Budgetary Healthcare Institution Saint - Petersburg, Saint Petersburg
  - Limited Liability Company "North-Western Medical Center", Saint Petersburg
  - Hospital OrKli LLC, Saint Petersburg
  - Federal State Budgetary Educational Institution of Higher Education, Saransk
  - Republican Clinical Oncology Dispensary of the Ministry of Health of Bashkortostan Republic, Ufa
  - Budgetary Healthcare Institution of Vologda region "Vologda Regional Clinical Hospital", Vologda
  - Leningrad Regional Clinical Hospital, Vsevolozhskiy District
  - SBHI YaR Regional clinical oncology hospital, Yaroslavl
- South Korea (7):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Kyungpook National University Chilgok Hospital, Daegu
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (19):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital General de Granollers, Granollers, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Salut Sant Joan de Reus-Baix Camp, Reus, Tarragona
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Hospital del Mar, Barcelona
  - Fundacio Puigvert, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital de Llíria, Llíria
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Fundacion Instituto Valenciano de Oncologia, Valencia
  - Hospital Arnau de Vilanova, Valencia
- United Kingdom (4):
  - Barts Health NHS Trust - St. Bartholomew's Hospital, London, CITY of London
  - Barts Health NHS Trust, of Royal London Hospital, London
  - Imperial College Healthcare NHS Trust, of The Bays, St. Mary's Hospital, London
  - Charing Cross Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Shore ND, Powles TB, Bedke J, Galsky MD, Palou Redorta J, Ku JH, Kretkowski M, Xylinas E, Alekseev B, Ye D, Guerrero-Ramos F, Briganti A, Kulkarni GS, Brinkmann J, Calella AM, Cesari R, Eccleston A, Michelon E, Vermette J, Wei C, Steinberg GD. Sasanlimab plus BCG in BCG-naive, high-risk non-muscle invasive bladder cancer: the randomized phase 3 CREST trial. Nat Med. 2025 Aug;31(8):2806-2814. doi: 10.1038/s41591-025-03738-z. Epub 2025 May 31. PMID 40450141
- [Derived] Steinberg GD, Shore ND, Redorta JP, Galsky MD, Bedke J, Ku JH, Kretkowski M, Hu H, Penkov K, Vermette JJ, Tarazi JC, Randall AE, Pierce KJ, Saltzstein D, Powles TB. CREST: phase III study of sasanlimab and Bacillus Calmette-Guerin for patients with Bacillus Calmette-Guerin-naive high-risk non-muscle-invasive bladder cancer. Future Oncol. 2024 May;20(14):891-901. doi: 10.2217/fon-2023-0271. Epub 2024 Jan 8. PMID 38189180
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B8011006

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in two cohorts: Cohort A (Bacillus Calmette Guerin [BCG] naïve participants with non-muscle invasive bladder cancer [NMIBC]) and Cohort B (BCG unresponsive participants with NMIBC).
Pre-assignment Details: A total of 1068 participants were enrolled in the study (Cohort A: 1055 participants, Cohort B1: 5 participants and Cohort B2: 8 participants). Results reported are based on the primary completion date (PCD) of the study; data for only those secondary outcome measures are reported for which analyses were complete at PCD. Remaining outcome measures would be reported upon completion of their analyses at study completion.
Groups:
- Cohort A, Arm A: PF-06801591+BCG (IND+MNT): Participants received PF-06801591 300 milligrams (mg) once every 4 weeks (Q4W) as a subcutaneous (SC) injection until Cycle 25. Full dose of BCG was administered as intravesical instillation once every week for 6 consecutive doses during Cycle 1 and Cycle 2 in the induction (IND) phase and on Days 1, 8 and 15 during Cycle 4, Cycle 7, Cycle 13, Cycle 19 and Cycle 25 in the maintenance (MNT) phase. For participants that had a re-induction period, the maintenance period started at C7D1 (1 cycle= 4 weeks).
- Cohort A, Arm B: PF-06801591+BCG (IND): Participants received PF-06801591 300 mg Q4W as a SC injection until Cycle 25. A full dose of BCG was administered as intravesical instillation once every week for 6 consecutive doses during Cycle 1 and Cycle 2 in the IND phase (1 cycle= 4 weeks).
- Cohort A, Arm C: BCG (IND+MNT): Participants were administered a full dose of BCG as intravesical instillation once every week for 6 consecutive doses during Cycle 1 and Cycle 2 in the IND phase and on Days 1, 8 and 15 during Cycle 4, Cycle 7, Cycle 13, Cycle 19 and Cycle 25 in the MNT phase. For participants that have a re-induction period, the maintenance period began at C7D1 (1 cycle= 4 weeks).
- Cohort B1: PF-06801591 300 mg: Participants with persistent or recurrent carcinoma in situ (CIS) alone or with concomitant recurrent Ta/T1 papillary disease received PF-06801591 300 mg Q4W as SC injection until Cycle 25 (1 cycle= 4 weeks).
- Cohort B2: PF-06801591 600 mg: Participants with high-grade Ta/T1 papillary disease received PF-06801591 600 mg once every 6 weeks (Q6W) as SC injection until Cycle 17 (1 cycle= 4 weeks).
Period: Treatment Phase
Arm/Group | Cohort A, Arm A: PF-06801591+BCG (IND+MNT) | Cohort A, Arm B: PF-06801591+BCG (IND) | Cohort A, Arm C: BCG (IND+MNT) | Cohort B1: PF-06801591 300 mg | Cohort B2: PF-06801591 600 mg
Started | 352 | 352 | 351 | 5 | 8
Treated | 350 | 348 | 349 | 5 | 8
Completed | 121 | 160 | 203 | 1 | 4
Not Completed | 231 | 192 | 148 | 4 | 4
Not completed — Adverse Event | 131 | 89 | 37 | 0 | 2
Not completed — Death | 8 | 8 | 6 | 0 | 0
Not completed — Lack of Efficacy | 32 | 50 | 54 | 3 | 2
Not completed — Lost to Follow-up | 3 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 41 | 26 | 29 | 1 | 0
Not completed — Global Deterioration of Health Status | 0 | 2 | 0 | 0 | 0
Not completed — Other | 14 | 13 | 18 | 0 | 0
Not completed — Randomized, not treated | 2 | 4 | 2 | 0 | 0
Period: Follow up Phase
Arm/Group | Cohort A, Arm A: PF-06801591+BCG (IND+MNT) | Cohort A, Arm B: PF-06801591+BCG (IND) | Cohort A, Arm C: BCG (IND+MNT) | Cohort B1: PF-06801591 300 mg | Cohort B2: PF-06801591 600 mg
Started | 319 (Participant who discontinued treatment could enter the follow up phase.) | 330 (Participant who discontinued treatment could enter the follow up phase.) | 334 (Participant who discontinued treatment could enter the follow up phase.) | 5 (Participant who discontinued treatment could enter the follow up phase.) | 7 (Participant who discontinued treatment could enter the follow up phase.)
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 319 | 330 | 334 | 5 | 7
Not completed — Death | 23 | 20 | 23 | 0 | 0
Not completed — Lost to Follow-up | 4 | 6 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 27 | 21 | 0 | 0
Not completed — Ongoing | 280 | 277 | 289 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 5 | 7

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) Cohort A included all participants who were randomized in Cohort A. For Cohort B1 and B2, Safety Analysis Set (SAS) was used which included all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A, Arm A: PF-06801591+BCG (IND+MNT) | Cohort A, Arm B: PF-06801591+BCG (IND) | Cohort A, Arm C: BCG (IND+MNT) | Cohort B1: PF-06801591 300 mg | Cohort B2: PF-06801591 600 mg | Total
Number analyzed (Participants) | 352 | 352 | 351 | 5 | 8 | 1068
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 142 | 141 | 133 | 2 | 3 | 421
  65 to <75 years | 135 | 141 | 142 | 1 | 2 | 421
  75 to <85 years | 71 | 62 | 66 | 2 | 3 | 204
  >=85 years | 4 | 8 | 10 | 0 | 0 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 53 | 67 | 0 | 0 | 192
  Male | 280 | 299 | 284 | 5 | 8 | 876
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 115 | 133 | 126 | 1 | 2 | 377
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 5 | 0 | 0 | 10
  White | 225 | 211 | 210 | 3 | 6 | 655
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 9 | 6 | 10 | 1 | 0 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino or of Spanish origin | 22 | 25 | 24 | 1 | 0 | 72
  Ethnicity: Not Hispanic or Latino or of Spanish origin | 315 | 314 | 310 | 3 | 8 | 950
  Ethnicity: Not Reported | 15 | 13 | 17 | 1 | 0 | 46

OUTCOME MEASURES:

1. Primary Outcome: Cohort A: Event Free Survival (EFS) as Assessed by the Investigator: Arm A Versus Arm C
Description: EFS: time from randomization till recurrence of high-grade disease, progression of disease, persistence of carcinoma in situ (CIS), death due to any cause, whichever occurred first. Recurrence of high-grade disease: re-appearance of high-grade disease after randomization/study intervention initiation, re-appearance of high-grade disease after complete response (CR) for CIS participants or re-appearance of high-grade disease before CR for CIS participants and concurrent papillary disease at baseline. Progression of disease defined as any of following: Lamina propria invasion, muscle invasive disease, lymph node positive disease, metastatic disease, high-grade stage of bladder cancer (non-invasive papillary carcinoma [Ta] or invasion into the lamina propria without invasion into the muscularis propria [T1]) in participants with CIS only at baseline before achieving CR. Persistence of CIS: persistent CIS after induction, re-induction. EFS estimated using Kaplan-Meier analysis.
Time Frame: From randomization (Day 1) to first documentation of high-grade disease, progression of disease, persistence of CIS or death due to any cause, whichever occurred first (maximum follow up duration was up to 257.1 weeks)
Population: Full analysis set (FAS) included all participants who were randomized in Cohort A.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A, Arm A: PF-06801591+BCG (IND+MNT) | Cohort A, Arm C: BCG (IND+MNT)
Number analyzed (Participants) | 352 | 351
Months | NA [NA to NA] — Median and 95% CI could not be estimated due to insufficient participants with events. | NA [NA to NA] — Median and 95% CI could not be estimated due to insufficient participants with events.
Statistical Analysis 1: Comparison: Cohort A, Arm A: PF-06801591+BCG (IND+MNT) vs Cohort A, Arm C: BCG (IND+MNT); Test type: Superiority; p = 0.0095, Log Rank; 1- sided p-value; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.489 to 0.941] — Hazard ratio was based on Cox proportional hazards model

2. Secondary Outcome: Cohort A: EFS as Assessed by the Investigator: Arm B Versus Arm C
Description: EFS: time from randomization till recurrence of high-grade disease, progression of disease, CIS, death due to any cause, whichever occurred first. Recurrence of high-grade disease: re-appearance of high-grade disease after randomization/study intervention initiation, re-appearance of high-grade disease after CR for CIS participants or re-appearance of high-grade disease before CR for CIS participants and concurrent papillary disease at baseline. Progression of disease defined as any of following: Lamina propria invasion, muscle invasive disease, lymph node positive disease, metastatic disease, high-grade stage of bladder cancer (non-invasive papillary carcinoma [Ta] or invasion into the lamina propria without invasion into the muscularis propria [T1]) in participants with CIS only at baseline before achieving CR. Persistence of CIS: persistent CIS after induction, re-induction. EFS estimated using Kaplan-Meier analysis.
Time Frame: From randomization (Day 1) to the first documentation of high-grade disease, progression of disease, persistence of CIS or death due to any cause, whichever occurred first (maximum follow up duration was up to 257.1 weeks)
Population: FAS included all participants who were randomized in Cohort A.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A, Arm B: PF-06801591+BCG (IND) | Cohort A, Arm C: BCG (IND+MNT)
Number analyzed (Participants) | 352 | 351
Months | 50.1 [47.1 to NA] — Upper limit of 95% CI could not be estimated due to insufficient participants with events. | NA [NA to NA] — Median and 95% CI could not be estimated due to insufficient participants with events.
Statistical Analysis 1: Comparison: Cohort A, Arm B: PF-06801591+BCG (IND) vs Cohort A, Arm C: BCG (IND+MNT); Test type: Superiority; p = 0.8439, Log Rank; 1 - sided p-value; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.870 to 1.552] — Hazard ratio was based on Cox proportional hazards model

3. Secondary Outcome: Cohort A: Overall Survival (OS) for Participants: Arm A Versus Arm C
Description: Overall survival was defined as the time in months from the date of randomization to the date of death due to any cause. Participants last known to be alive will be censored at the date of last contact
Time Frame: From randomization (Day 1) until date of death due to any cause or censoring date
Reporting Status: Not Posted, anticipated posting 2027-12

4. Secondary Outcome: Cohort A: OS of Participants: Arm B Versus Arm C
Description: as for outcome 3
Time Frame: From randomization (Day 1) until date of death due to any cause or censoring date
Reporting Status: Not Posted, anticipated posting 2027-12

5. Secondary Outcome: Cohort A: Percentage of Participants With Complete Response (CR)as Assessed by Investigator: Participants With CIS at Baseline in Full Analysis Set
Description: CR was defined as histologic disappearance of malignancy on bladder biopsy with negative cytology and cystoscopy or negative cytology and positive cystoscopy with biopsy-proven low-grade stage of bladder cancer defined as a non-invasive papillary carcinoma (Ta) lesion or non-malignant tissue for participants with CIS at randomization. 95% CI was based on Clopper-Pearson method.
Time Frame: From randomization (Day 1) to the first documented CR (maximum follow up duration was up to 257.1 weeks)
Population: FAS included all participants who were randomized in Cohort A. Here, "Overall Number of Participants Analyzed" (N) signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A, Arm A: PF-06801591+BCG (IND+MNT) | Cohort A, Arm B: PF-06801591+BCG (IND) | Cohort A, Arm C: BCG (IND+MNT)
Number analyzed (Participants) | 88 | 93 | 88
Percentage of participants | 89.8 [81.5 to 95.2] | 88.2 [79.8 to 93.9] | 85.2 [76.1 to 91.9]

6. Secondary Outcome: Cohort A: Duration of CR as Assessed by the Investigator: Participants With CIS at Baseline in Full Analysis Set
Description: Duration of CR was defined as the time from the first documentation of CR to the date of an EFS event for participants with CR. EFS was defined as the time in months from randomization until recurrence of high-grade disease, progression of disease, persistence of CIS or death due to any cause, whichever occurred first. CR was defined as histologic disappearance of malignancy on bladder biopsy with negative cytology and cystoscopy or negative cytology and positive cystoscopy with biopsy-proven low-grade stage of bladder cancer defined as a non-invasive papillary carcinoma (Ta) lesion or non-malignant tissue for participants with CIS at randomization. Kaplan-Meier method was used. 95% CI was estimated based on Brookmeyer and Crowley method.
Time Frame: From date of first documentation of CR to date of an EFS event (maximum follow up duration was up to 257.1 weeks)
Population: FAS included all participants who were randomized in Cohort A. Here, "Overall Number of Participants Analyzed" included the participants with CIS at Baseline from FAS who achieved CR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A, Arm A: PF-06801591+BCG (IND+MNT) | Cohort A, Arm B: PF-06801591+BCG (IND) | Cohort A, Arm C: BCG (IND+MNT)
Number analyzed (Participants) | 79 | 82 | 75
Months | NA [NA to NA] — Median and 95% CI could not be estimated due to insufficient participants with events. | 44.6 [44.6 to NA] — Upper limit for 95% CI could not be estimated due to insufficient participants with events. | NA [39.3 to NA] — Median and upper limit for 95% CI could not be estimated due to insufficient participants with events.

7. Secondary Outcome: Cohort A: Time to Recurrence of Low-Grade Disease Assessed by the Investigator
Description: Time to recurrence of low-grade disease was defined as the time from randomization to the date of first documentation of recurrence of low-grade disease. Recurrence of low-grade disease was defined as re-appearance of low-grade disease (low-grade Ta) after randomization based on positive biopsy, cystoscopy or cytology result. Kaplan-Meier method was used. 95% CI was estimated based on Brookmeyer and Crowley method.
Time Frame: From randomization (Day 1) to the date of positive biopsy, cystoscopy or cytology results (maximum follow up duration was up to 257.1 weeks)
Population: FAS included all participants who were randomized in Cohort A.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A, Arm A: PF-06801591+BCG (IND+MNT) | Cohort A, Arm B: PF-06801591+BCG (IND) | Cohort A, Arm C: BCG (IND+MNT)
Number analyzed (Participants) | 352 | 352 | 351
Months | 48.8 [NA to NA] — 95% CI for Arm A could not be estimated due to insufficient participants with events, and the lower limit of the 95% confidence interval could not be calculated due to heavy censoring prior to the last participant having an event. | NA [47.9 to NA] — Median and upper limit for 95% CI could not be estimated due to insufficient participants with events. | NA [NA to NA] — Median and 95% CI could not be estimated due to insufficient participants with events.

8. Secondary Outcome: Cohort A: Time to Cystectomy
Description: Time to cystectomy was defined as time from randomization to cystectomy. Participants without a cystectomy will be censored at death date or last date known to be alive.
Time Frame: From randomization (Day 1) to date of cystectomy or censoring date
Population: Intent-to-treat (ITT) Population: all randomized participants
Reporting Status: Not Posted, anticipated posting 2027-12

9. Secondary Outcome: Cohort A: Disease Specific Survival (DSS) as Assessed by the Investigator
Description: DSS was defined as the time from randomization to death resulting from bladder cancer, as assessed by the investigator. Participants last known to be alive will be censored at the date of last contact.
Time Frame: From randomization (Day 1) to the first documentation of death from bladder cancer
Population: Intent-to-treat (ITT) Population: all randomized participants
Reporting Status: Not Posted, anticipated posting 2027-12

10. Secondary Outcome: Cohort A: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. TEAEs were those events with onset dates occurring during the on-treatment period. On-treatment period was defined as the time from the first dose of study treatment up to 30 days after last dose of study treatment or 1 day before start day of new anti-cancer therapy.
Time Frame: From first dose of study treatment (Day 1) up to 30 days after last dose of study treatment or 1 day before anti-cancer therapy
Reporting Status: Not Posted, anticipated posting 2027-12

11. Secondary Outcome: Cohort A: Number of Participants With Serious TEAEs
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. TEAEs were those events with onset dates occurring during the on-treatment period. On-treatment period was defined as the time from the first dose of study treatment up to 30 days after last dose of study treatment or 1 day before start day of new anti-cancer therapy. A serious adverse event (SAE) was any untoward medical occurrence at any dose that: resulted in death or was life threatening or required inpatient hospitalization or prolongation of existing hospitalization or resulted in persistent or significant disability/incapacity, resulted in congenital anomaly/birth defect or other events.
Time Frame: as for outcome 10
Reporting Status: Not Posted, anticipated posting 2027-12

12. Secondary Outcome: Cohort A: Number of Participants With Treatment Related TEAEs and Treatment Related SAEs
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. TEAEs were those events with onset dates occurring during the on-treatment period. On-treatment period was defined as the time from the first dose of study treatment up to 30 days after last dose of study treatment or 1 day before start day of new anti-cancer therapy. A SAE was any untoward medical occurrence at any dose that: resulted in death or was life threatening or required inpatient hospitalization or prolongation of existing hospitalization or resulted in persistent or significant disability/incapacity resulted in congenital anomaly/birth defect or other events. Relatedness was based on the investigator's judgement.
Time Frame: as for outcome 10
Reporting Status: Not Posted, anticipated posting 2027-12

13. Secondary Outcome: Cohort A: Number of Participant With Grade 3 or 4 and Grade 5 TEAEs Based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. TEAEs were those events with onset dates occurring during the on-treatment period. On-treatment period was defined as the time from the first dose of study treatment up to 30 days after last dose of study treatment or 1 day before start day of new anti-cancer therapy. NCI-CTCAE version 5.0, severity was graded as Grade 1: Mild, Grade 2: Moderate, Grade 3: Severe and Grade 4 Life threatening and Grade 5: Death.
Time Frame: as for outcome 10
Reporting Status: Not Posted, anticipated posting 2027-12

14. Secondary Outcome: Cohort A: Number of Participant With Laboratory Abnormalities as Based on Severity (as Graded by NCI CTCAE v5.0)
Description: Laboratory parameters: hematocrit, hemoglobin, platelets, white blood cells, absolute neutrophil count, lymphocytes, monocytes, eosinophils, basophils, alanine aminotransferase, aspartate aminotransferase, lactate dehydrogenase, alkaline phosphatase, sodium, potassium, magnesium, chloride, total calcium and bilirubin, blood urea nitrogen, urea, creatinine, uric acid, glucose (non-fasted), albumin, phosphorus/phosphate, lipase, amylase, thyroid function test + reflex free thyroxine, free triiodothyronine, adrenocorticotropic hormone, international normalized ratio, partial thromboplastin time (PTT)/activated PTT, hepatitis B surface antigen, hepatitis C virus antibody. Severity grades per NCI-CTCAE v5.0: 1: Mild, 2: Moderate, 3: Severe, 4: Life threatening,5: Death.
Time Frame: as for outcome 10
Reporting Status: Not Posted, anticipated posting 2027-12

15. Secondary Outcome: Cohort A: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Non-Muscle Invasive Bladder Cancer (QLQ-C) 30 Total Score
Description: The EORTC QLQ-C30 was a 30 self-administered questionnaire, which comprised of 5 functional domain subscales (physical functioning subscale, a role functioning subscale, an emotional functioning subscale, a cognitive functioning subscale and a social functioning subscale), 3 symptom scale (fatigue, pain, nausea and vomiting), 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial impact) and a global health status/QoL scale. All the scales and single-item measures range in score from 0 (poor functioning/no symptoms) to 100 (excellent functioning/greater degree of symptoms). Higher scores on functional domains indicated higher levels of functioning and higher scores on symptom scale/single items indicated greater presence of symptoms.
Time Frame: Baseline up to recurrence of high-grade disease or disease progression, consent withdrawal, lost to follow-up, or death
Reporting Status: Not Posted, anticipated posting 2027-12

16. Secondary Outcome: Cohort A: Change From Baseline in EORTC QLQ- Non-Muscle Invasive Bladder Cancer (NMIBC24) Total Score
Description: The EORTC QLQ NMIBC24 is a PRO developed and tested by the EORTC group specifically for participants with non-muscle invasive bladder cancer. The NMIBC24 has 24 items which can be grouped into 6 subscales: urinary symptoms (7 items), malaise (2 items), future worries (4 items), bloating/flatulence (2 items), sexual functioning (2 items), and male sexual issues (2 items). The NMIBC24 also assesses intravesical treatment, female sexual issues, sexual intimacy, risk of contaminating a partner, and sexual enjoyment (1 item each). All of the subscales and single-item measures range in score from 0 (poor functioning/no symptoms) to 100 (excellent functioning/greater degree of symptoms). Higher scores indicate greater impairment, except for sexual function and sexual enjoyment items, where higher scores indicate better function.
Time Frame: Baseline up to recurrence of high-grade disease or disease progression, consent withdrawal, lost to follow-up, or death
Reporting Status: Not Posted, anticipated posting 2027-12

17. Secondary Outcome: Cohort A: Change From Baseline in Patient Treatment Administration Burden (PTAB) Questionnaire Total Score
Description: The PTAB questionnaire was a 2-item PRO designed to assess, from the participant perspective, any pain associated with the treatment administration and the burden of the amount of time required to complete the treatment administration procedures (1 item each). The items were scored on a range of 0 to 4, where 0=no pain/ not at all burdensome and 4= extremely severe pain/ extremely burdensome.
Time Frame: Baseline up to 7 days after last dose of study treatment
Reporting Status: Not Posted, anticipated posting 2027-12

18. Secondary Outcome: Cohort A: Concentration at Trough (Ctrough) of PF-06801591 for Arms A and B Only
Description: Concentration at Trough is defined as Predose/trough concentration Observed directly from data.
Time Frame: Pre-dose on Day 1 of Cycles 1, 2, 4, 6, 8, 10 and 13 (1 cycle=4 weeks)
Population: PK concentration analysis set =subset of safety analysis set and included participants who had at least one post-dose concentration measurement above lower limit of quantitation (LLOQ) for PF-06801591. "Overall Number of Participants Analyzed"=participants evaluable for this outcome measure and "Number Analyzed" =participants evaluable for specific row. This outcome measure was planned to be analyzed only for PF-06801591 as pre-specified in the protocol; hence, only Arm A and B are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Cohort A, Arm A: PF-06801591+BCG (IND+MNT) | Cohort A, Arm B: PF-06801591+BCG (IND)
Number analyzed (Participants) | 315 | 314
Nanogram per milliliter (ng/mL)
  Cycle 1 (Day 1): number analyzed (Participants) | 315 | 1
  Cycle 1 (Day 1) | NA [NA to NA] — Geometric mean and 95 % Confidence interval could not be estimated as the values were below the lower limit of quantification (LLOQ). | NA [NA to NA] — Geometric mean and 95 % Confidence interval could not be estimated as the values were below the lower limit of quantification.
  Cycle 2 (Day1): number analyzed (Participants) | 313 | 314
  Cycle 2 (Day1) | 17530.0 [16848.8 to 18238.8] | 17398.8 [16569.0 to 18270.0]
  Cycle 4 (Day1): number analyzed (Participants) | 237 | 255
  Cycle 4 (Day1) | 30587.9 [29256.1 to 31980.4] | 30507.1 [29043.6 to 32044.3]
  Cycle 6 (Day 1): number analyzed (Participants) | 220 | 223
  Cycle 6 (Day 1) | 32945.2 [31352.8 to 34618.5] | 34614.0 [32634.8 to 36713.2]
  Cycle 8 (Day 1): number analyzed (Participants) | 187 | 201
  Cycle 8 (Day 1) | 35701.1 [34030.3 to 37454.0] | 36414.1 [33579.4 to 39488.1]
  Cycle 10 (Day 1): number analyzed (Participants) | 177 | 196
  Cycle 10 (Day 1) | 38616.9 [36395.7 to 40973.6] | 38965.4 [36374.5 to 41740.9]
  Cycle 13 (Day 1): number analyzed (Participants) | 153 | 153
  Cycle 13 (Day 1) | 41969.4 [39420.4 to 44683.3] | 41737.1 [39045.7 to 44614.1]

19. Secondary Outcome: Cohort A: Number of Participants With Positive (Anti-Drug Antibody) ADA or (Neutralizing Antibody) NAb: Arms A and B Only
Description: A participant was considered ADA (or NAb) positive if (1) baseline titer was missing or negative and participant had >= 1 post-treatment positive titer (treatment-induced), or (2) positive titer at baseline and had a >= 4-fold dilution increase in titer from baseline in >= 1 post-treatment sample (treatment-boosted).
Time Frame: From start of study treatment (Day 1) until 7 days after last dose of study treatment (maximum up to 125.1 weeks and 104.4 weeks of treatment exposure for Arm A and Arm B, respectively)
Population: Immunogenicity analyses set was subset of the safety population and included participants who received at least one dose of PF-06801591 and had at least one ADA/Nab sample analyzed for anti-PF-06801591 antibodies. "Overall Number of Participants Analyzed" =participants evaluable for this outcome measure" set. This outcome measure was planned to be analyzed only for PF-06801591 as pre-specified in the protocol; hence, only Arm A and B are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A, Arm A: PF-06801591+BCG (IND+MNT) | Cohort A, Arm B: PF-06801591+BCG (IND)
Number analyzed (Participants) | 345 | 343
Participants
  ADA | 19 | 19
  NAb | 0 | 1

20. Secondary Outcome: Cohort A: Number of Participants According to Tumor Sample Biomarker Status Based on Baseline Programmed Cell Death Ligand 1 (PD-L1) Expression
Description: PD-L1 expression was defined as the number of PD-L1 positive cells and/or qualitative assessment of PD-L1 staining on tumor and immune cells in regions of interest that were defined by tumor cell morphology. PDL-1 status was high if >=25% tumor cell or (immune cells present in the tumor area > 1% and PD-L1 positive immune cells+ >=25%) or (immune cells present in the tumor area = 1% and PD-L1 positive immune cells = 100%), and low if < 25% tumor cell and [(immune cells present in the tumor area > 1% and immune cells <25%) or (immune cells present in the tumor area = 1% and PD-L1 positive immune cells< 100%) or immune cells present = 0].
Time Frame: From start of study treatment (Day 1) until 7 days after last dose of study treatment (maximum up to 125.1 weeks, 104.4 weeks and 110 weeks of treatment exposure for Arm A, Arm B and Arm C, respectively)
Population: The biomarker analyses set were a subset of the safety population and included participants with at least 1 of the biomarkers evaluated at pre and/or post dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A, Arm A: PF-06801591+BCG (IND+MNT) | Cohort A, Arm B: PF-06801591+BCG (IND) | Cohort A, Arm C: BCG (IND+MNT)
Number analyzed (Participants) | 340 | 337 | 337
Participants
  High | 77 | 68 | 73
  Low | 252 | 256 | 253
  Unknown | 11 | 13 | 11

ADVERSE EVENTS:
Time Frame: From first dose of study treatment (Day 1) up to 30 days after last dose of study treatment or 1 day before anti-cancer therapy (maximum follow up duration was up to 257.1 weeks)
Description: Same event may appear as both non-serious adverse event and serious adverse event (SAE); however, what is presented are distinct events. Event may be categorized as serious in 1 participant and non-serious in another or 1 participant may have experienced both SAE and non-SAE. SAS included all participants who received at least 1 dose of study drug. All-cause mortality have been reported for full analysis set.
Arm/Group | Cohort A, Arm A: PF-06801591+BCG (IND+MNT) | Cohort A, Arm B: PF-06801591+BCG (IND) | Cohort A, Arm C: BCG (IND+MNT) | Cohort B1: PF-06801591 300 mg | Cohort B2: PF-06801591 600 mg
All-Cause Mortality (participants affected / at risk) | 32/352 | 30/352 | 29/351 | 0/5 | 0/8
Serious Adverse Events (participants affected / at risk) | 120/350 | 99/348 | 49/349 | 2/5 | 2/8
Other Adverse Events (participants affected / at risk) | 321/350 | 299/348 | 287/349 | 5/5 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A, Arm A: PF-06801591+BCG (IND+MNT) (N=350) | Cohort A, Arm B: PF-06801591+BCG (IND) (N=348) | Cohort A, Arm C: BCG (IND+MNT) (N=349) | Cohort B1: PF-06801591 300 mg (N=5) | Cohort B2: PF-06801591 600 mg (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 1 | 0 | 0
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 1 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Bundle branch block right (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 2 | 0 | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 3 | 0 | 1 | 0 | 0
Immune-mediated myocarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 3 | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 2 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0
Otolithiasis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 3 | 3 | 0 | 0 | 0
Hypophysitis (Endocrine disorders) | 1 | 1 | 0 | 1 | 0
Hypopituitarism (Endocrine disorders) | 2 | 2 | 0 | 0 | 0
Hypothalamo-pituitary disorder (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Immune-mediated hypophysitis (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Lymphocytic hypophysitis (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Secondary adrenocortical insufficiency (Endocrine disorders) | 1 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 1 | 0 | 0 | 0
Diabetic retinopathy (Eye disorders) | 1 | 0 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0 | 0 | 0
Uveitis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Intestinal mass (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Lymphocytic oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 4 | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 2 | 1 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 2 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0 | 0
Vascular stent stenosis (General disorders) | 1 | 0 | 0 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cholestatic liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Immune-mediated hepatic disorder (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 6 | 5 | 4 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 3 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Disseminated Bacillus Calmette-Guerin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Epididymitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Myringitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Orchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Otitis media chronic (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Parotitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 9 | 3 | 4 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Prostatitis tuberculous (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pyelonephritis chronic (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 0 | 0
Sepsis (Infections and infestations) | 4 | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Suspected COVID-19 (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 5 | 1 | 1 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Rectal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Urethral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood osmolarity decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 0 | 0
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Autoimmune myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Oligoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 0 | 0
Cardiac valve fibroelastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Hepatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0 | 0
Cerebellar stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 2 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Lacunar infarction (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Myasthenic syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Alcoholism (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 4 | 0 | 0 | 0
Calculus urethral (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Cystitis interstitial (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Diabetic nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Glomerulonephritis membranous (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Nephritis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Aneurysm (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Aortic dissection (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Arterial insufficiency (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Cyanosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Embolism arterial (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Giant cell arteritis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Haemorrhagic vasculitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 0 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A, Arm A: PF-06801591+BCG (IND+MNT) (N=350) | Cohort A, Arm B: PF-06801591+BCG (IND) (N=348) | Cohort A, Arm C: BCG (IND+MNT) (N=349) | Cohort B1: PF-06801591 300 mg (N=5) | Cohort B2: PF-06801591 600 mg (N=8)
Anaemia (Blood and lymphatic system disorders) | 27 | 27 | 13 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 30 | 29 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 55 | 49 | 3 | 1 | 1
Constipation (Gastrointestinal disorders) | 41 | 25 | 21 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 41 | 39 | 19 | 1 | 0
Nausea (Gastrointestinal disorders) | 25 | 11 | 11 | 0 | 0
Asthenia (General disorders) | 39 | 33 | 20 | 0 | 0
Fatigue (General disorders) | 52 | 42 | 21 | 1 | 2
Pyrexia (General disorders) | 74 | 51 | 52 | 1 | 0
COVID-19 (Infections and infestations) | 28 | 20 | 23 | 1 | 0
Cystitis (Infections and infestations) | 43 | 18 | 37 | 0 | 0
Urinary tract infection (Infections and infestations) | 90 | 54 | 82 | 0 | 2
Alanine aminotransferase increased (Investigations) | 56 | 38 | 30 | 2 | 0
Amylase increased (Investigations) | 56 | 42 | 15 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 53 | 37 | 25 | 0 | 0
Blood creatinine increased (Investigations) | 31 | 23 | 10 | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 23 | 14 | 10 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 7 | 19 | 3 | 0 | 0
Lipase increased (Investigations) | 76 | 56 | 28 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 56 | 37 | 49 | 0 | 0
Weight decreased (Investigations) | 32 | 17 | 9 | 0 | 1
Weight increased (Investigations) | 14 | 13 | 22 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 30 | 35 | 3 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 20 | 24 | 17 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 20 | 12 | 22 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 52 | 43 | 14 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 23 | 22 | 16 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 18 | 16 | 8 | 0 | 0
Headache (Nervous system disorders) | 29 | 20 | 14 | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 16 | 11 | 21 | 0 | 0
Dysuria (Renal and urinary disorders) | 115 | 72 | 126 | 2 | 0
Haematuria (Renal and urinary disorders) | 97 | 51 | 90 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 40 | 16 | 41 | 1 | 0
Nocturia (Renal and urinary disorders) | 20 | 7 | 20 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 83 | 39 | 74 | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 18 | 10 | 17 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 23 | 12 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 14 | 7 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 48 | 43 | 8 | 1 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 21 | 11 | 2 | 0 | 0
Hypertension (Vascular disorders) | 22 | 24 | 33 | 1 | 0
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Urethral pain (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Arterial disorder (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Bladder perforation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Enrollment in Cohort B was closed based on sponsors decision; hence, the study objectives for Cohorts B1 and B2 were no longer required as pre-specified in the protocol; outcome measures for Cohorts B based on the data collected will be summarized and reported at the time of final analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2024-06-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT04165317/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT04165317/SAP_001.pdf